CLINICAL TRIAL: NCT04666662
Title: Development and Validation of a Prognostic Model to PREDICT Relapse of Depression in Adult Patients in Primary Care
Brief Title: A Prognostic Model to PREDICT Relapse of Depression in Primary Care
Acronym: PREDICTR
Status: Completed | Type: Observational
Sponsor: University of York (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); Keele University (Other)
Responsible Party: Principal Investigator, Andrew Moriarty, NIHR Doctoral Research Fellow, University of York
Other Study IDs: 11ST2044
Record Dates: First submitted 2020-12-07; First posted 2020-12-14 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Depression
Keywords: Prediction; Prognostic model; Relapse
MeSH Terms: conditions — Depression; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators aim to develop a prognostic model to predict the risk of relapse within 6-8 months of patients entering remission. The long-term objective is to facilitate more efficient targeting of evidence-based relapse prevention strategies to these patients.

DETAILED DESCRIPTION:
Most patients with depression are treated in primary care by general practitioners (GPs). Relapse of depression is common and leads to considerable morbidity and decreased quality of life for patients. Estimates suggest that at least 50% of patients treated for depression will relapse after a single episode. The majority of these will relapse within 6 months and the risk of relapse increases for each successive episode of depression. GPs see a largely undifferentiated case-mix of patients and, once patients with depression reach remission, there is limited guidance and no validated tools to help GPs stratify patients according to risk of relapse.This study will potentially derive a statistical model to predict relapse of depression in remitted depressed patients in primary care.

The investigators have created a longitudinal cohort of patients drawn from seven randomised controlled trials (RCTs) of non-pharmacological primary care-based interventions for depression and one longitudinal cohort study. The investigators will use logistic regression to predict the outcome of relapse of depression within 6-8 months. The investigators plan to include the following well-evidenced relapse predictors in the model: residual depressive symptoms; number of previous episodes of depression; co-morbid anxiety; and severity of the index episode. They will also control for RCT intervention received by participants.

If sample size and availability of predictor information allows, the investigators will include the following predictors in an exploratory analysis: age; relationship status; multi-morbidity; employment status; gender; and ethnicity. Generalisability will be assessed through internal-external cross-validation and net benefit will be explored.

ELIGIBILITY:
Inclusion Criteria:

* Remitted depressive disorder

Exclusion Criteria:

* Co-existing severe mental illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will represent an undifferentiated primary care case-mix of patients with depression, meeting clinical criteria for remission at the point of prediction.
Sampling Method: Non-Probability Sample
Enrollment: 1244 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2024-06-24 (Actual); Study Completion 2024-06-24 (Actual)

PRIMARY OUTCOMES:
Whether a participant relapses or not within 6-8 months (binary outcome) | 6-8 months
  Relapse is the re-emergence of depressive symptoms according to Patient Health Questionnaire (PHQ-9)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Moriarty, MRes, Principal Investigator — University of York
Locations (1):
- University of York, York, United Kingdom

REFERENCES:
- [Derived] Moriarty AS, Paton LW, Snell KIE, Archer L, Riley RD, Buckman JEJ, Chew Graham CA, Gilbody S, Ali S, Pilling S, Meader N, Phillips B, Coventry PA, Delgadillo J, Richards DA, Salisbury C, McMillan D. Development and validation of a prognostic model to predict relapse in adults with remitted depression in primary care: secondary analysis of pooled individual participant data from multiple studies. BMJ Ment Health. 2024 Oct 28;27(1):e301226. doi: 10.1136/bmjment-2024-301226. PMID 39467616
- [Derived] Moriarty AS, Paton LW, Snell KIE, Riley RD, Buckman JEJ, Gilbody S, Chew-Graham CA, Ali S, Pilling S, Meader N, Phillips B, Coventry PA, Delgadillo J, Richards DA, Salisbury C, McMillan D. The development and validation of a prognostic model to PREDICT Relapse of depression in adult patients in primary care: protocol for the PREDICTR study. Diagn Progn Res. 2021 Jul 2;5(1):12. doi: 10.1186/s41512-021-00101-x. PMID 34215317